CLINICAL TRIAL: NCT01141270
Title: Comparative Pharmacokinetics of AFOLIA and Gonal-f® After Single Subcutaneous Application. A Randomised, Open Label, Cross Over Study
Brief Title: Comparative Pharmacokinetics of AFOLIA and Gonal-f® After Single Subcutaneous Application
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Polymun Scientific GmbH (Industry)
Responsible Party: Brigitta Vcelar PhD, Polymun Scientific GmbH
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: FIN1001
Record Dates: First submitted 2010-06-09; First posted 2010-06-10 (Estimated); Last update posted 2010-08-04 (Estimated); Status verified 2010-08

CONDITIONS: Healthy
Keywords: recombinant human follicle stimulating hormone; pharmacokinetics; bioequivalence
MeSH Terms: interventions — follitropin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AFOLIA (Experimental): 225 IU sc
  Interventions: Drug: AFOLIA
- Gonal-f (Active Comparator): 225 IU sc
  Interventions: Drug: Gonal-f

INTERVENTIONS:
Drug: AFOLIA — single sc injection, 225 IU
  Arms: AFOLIA
Drug: Gonal-f — single sc injection, 225IU
  Arms: Gonal-f

SUMMARY:
Comparative pharmacokinetics study after single subcutaneous application of AFOLIA and the reference product (Gonal-f®).

Objective: To demonstrate equivalence within the 80%-125% margin of the reference product for the area under the curve (AUC) of AFOLIA compared to (Gonal-f®).

ELIGIBILITY:
Inclusion Criteria:

* Healthy female volunteers
* Age between 18-38 years
* Body mass index 17-29 kg/m2
* Woman of child bearing potential must agree to practice effective barrier methods for birth control
* Use of oral contraceptives for at least 3 months before study entry
* Regular menstruation cycle (25-34 days) before initiation of oral contraception
* Presence of both ovaries
* Normal findings in medical history and physical and gynaecological examination unless the investigator considers an abnormality to be clinically irrelevant for this study
* Signed informed consent

Exclusion Criteria:

* Polycystic ovary syndrome (PCOS)
* History of hypersensitivity to FSH (Ovary Hyperstimulation Syndrome, OHSS)
* Impaired thyroid function (treated or untreated)
* History of malignant disease
* AST and/or ALAT > 2 x ULN
* Other clinically relevant findings (ECG, blood pressure, physical, gynecological examination, laboratory examination)
* Smoking habits of more than 5 cigarettes per day
* Abuse of alcoholic beverages and drugs
* Participation in a clinical trial within 3 weeks prior to the study
* Foreseen inability to attend to scheduled study visits
* Symptoms of a clinically relevant illness during 3 weeks prior the first study day
* Pregnancy or lactation period
* Any medical condition that, in the opinion of the investigator, would interfere with safety of the subject or interference of the objectives of the study

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2009-01; Primary Completion 2009-08 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Area under the serum concentration curve (AUC) of FSH | 0 -192h after FSH injection

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wolzt, aoUniv.Prof., Principal Investigator — Medical University Vienna